CLINICAL TRIAL: NCT01512966
Title: An Open-label Phase III Study Evaluating the Safety and Tolerability of Repeated Doses of Intravitreal VEGF Trap-Eye in Japanese Subjects With Diabetic Macular Edema
Brief Title: Japanese Safety Study of VEGF Trap-Eye in DME (Diabetic Macular Edema)
Acronym: VIVID-Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15657
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Macular Edema
Keywords: Diabetic Macular Edema; DME; VEGF Trap-Eye; best-corrected visual acuity (BCVA)
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VTE 2Q4 first, then VTE 2Q8 (Experimental): VEGF Trap-Eye [BAY86-5321; EYLEA (aflibercept) Injection] 2 mg Q4 (VTE 2Q4) administered every 4 weeks from Week 0 to Week 16, followed by every 8 weeks until Week 48 (2Q8)
  Interventions: Biological: VEGF Trap-Eye (BAY86-5321)

INTERVENTIONS:
Biological: VEGF Trap-Eye (BAY86-5321) — Subjects in the VEGF Trap-Eye group will receive intravitreal injections every 8 weeks following a loading phase with injections given every 4 weeks. The overall treatment period is 48 weeks.

SUMMARY:
This study will assess the safety and tolerability of intravitreally (IVT) administered VEGF Trap-Eye in Japanese subjects with diabetic macular edema (DME) over the period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus
* Subjects with DME (diabetic macular edema) secondary to diabetes mellitus involving the center of the macula in the study eye
* BCVA (best-corrected visual acuity) ETDRS (Early Treatment Diabetic Retinopathy Study) letter score of 73 to 24 (20/40 to 20/320) in the study eye

Exclusion Criteria:

* Active proliferative diabetic retinopathy (PDR) in the study eye
* Uncontrolled diabetes mellitus, as defined by HbA1c >12%
* Only 1 functional eye even if that eye is otherwise eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Adverse Event collection | Week 52

SECONDARY OUTCOMES:
Change from baseline in BCVA (best corrected visual acuity) letter score | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Japan (17):
  - Matsuyama, Ehime
  - Maebashi, Gunma
  - Kobe, Hyōgo
  - Mito, Ibaraki
  - Kita, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kawasaki, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Kashihara, Nara
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Suita, Osaka
  - Saga, Saga-ken
  - Ōtsu, Shiga
  - Shimotsuke, Tochigi
  - Wakayama, Wakayama